CLINICAL TRIAL: NCT05349201
Title: CAR-T Cells - Real Life Study Of Care Pathway And Total Cost Of Care For Patients Under Car T-Cell Treatment Based On The PMSI French Database
Brief Title: CAR T Cells Real World Evidence Study Based on the French Hospital Claims Data Source (PMSI)
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CCTL019A0FR02
Record Dates: First submitted 2022-04-06; First posted 2022-04-27 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Diffuse Large B-Cell Lymphoma (DLBCL); Acute Lymphoblastic Leukemia (ALL)
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — tisagenlecleucel; axicabtagene ciloleucel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- Adult R/R DLBCL cohort: KYMRIAH: Patients (≥18 years of age) with (relapsed/refractory diffuse large B cell lymphoma [R/R DLBCL])
  Interventions: Other: KYMRIAH
- Adult R/R DLBCL cohort: YESCARTA: Patients (≥18 years of age) with (relapsed/refractory diffuse large B cell lymphoma [R/R DLBCL])
  Interventions: Other: YESCARTA
- ALL pediatric and young adult cohort: KYMRIAH: Pediatric and young adult patients (≤25 years of age) with B cell acute lymphoblastic leukemia (ALL) ( refractory, in relapse post transplant or in second or later relapse
  Interventions: Other: KYMRIAH

INTERVENTIONS:
Other: KYMRIAH — Patients (≥18 years of age) with (relapsed/refractory diffuse large B cell lymphoma [R/R DLBCL]) or Pediatric and young adult patients (≤25 years of age) with B cell acute lymphoblastic leukemia (ALL) refractory, in relapse post transplant or in second or later relapse
  Groups: ALL pediatric and young adult cohort: KYMRIAH; Adult R/R DLBCL cohort: KYMRIAH
Other: YESCARTA — Patients (≥18 years of age) with (relapsed/refractory diffuse large B cell lymphoma [R/R DLBCL])
  Groups: Adult R/R DLBCL cohort: YESCARTA

SUMMARY:
This was a Retrospective cohort study based on the PMSI data source

DETAILED DESCRIPTION:
A retrospective database analysis was performed using the French national hospital claims database (Medicalized Information System Program - PMSI, 2015-2019), which includes discharge summaries for all hospital admissions in France (~99% of French residents).

The patients were identified based on the CAR-T administration hospital stay, between 2017 and 2019. Based on the exhaustivity of the database, all patients treated with CAR-T (since 2018) were identified.

The study design included multiple periods of analysis based on the CAR-T process. Three main periods were defined: the historical period, the CAR-T period, and the post CAR-T period. The CAR-T period was divided in 2 sub-periods: pre CAR-T (including the apheresis procedure and 15 days before this procedure) and per CAR-T (including the lymphodepletion and CAR-T cell injection hospital stay until the end at the discharge date related to CAR-T cell injection hospital stay). The follow-up period started at the end of CAR-T hospital stay.

CAR-T populations:

KYMRIAH® DLBCL cohort:

* Adult patients (≥18 years of age) with relapsed or refractory diffuse large B-cell lymphoma (DLBCL) after two or more lines of systemic therapy.
* Patient with a CAR-T administration hospital stay of Kymriah between 2017 and 2019

YESCARTA®DLBCL cohort:

* Adult patients (≥18 years of age) with relapsed or refractory diffuse large B-cell lymphoma (DLBCL) after two or more lines of systemic therapy:
* Patient with a CAR-T administration hospital stay of Yescarta between 2017 and 2019

KYMRIAH® ALL cohort:

* Pediatric and young adult patients (≤ 25 years of age) with B-cell acute lymphoblastic leukemia (ALL) that is refractory, in relapse post-transplant or in second or later relapse:
* Patient with a CAR-T administration hospital stay of Kymriah between 2017 and 2019

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with CAR-T cells from 2017 to 2019 and informed as such in the PMSI And
* Patients diagnosed with ALL or DLBCL when administering CAR-T cells and
* up to 25 years for patients with ALL

Exclusion Criteria:

* All patients treated outside the two types of indications presented in the inclusion criteria will be excluded

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients ( ≥18 years of age) with (relapsed/refractory diffuse large B cell lymphoma [R/R DLBCL]), currently being treated in third line or more with
  * KYMRIAH
  * YESCARTA
  Pediatric and young adult patients (≤25 years of age) with B cell acute lymphoblastic leukemia ( refractory, in relapse post transplant or in second or later relapse, currently being treated in third line or higher with
  • KYMRIAH
Sampling Method: Non-Probability Sample
Enrollment: 273 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
Overall survival: number of events | through study completion, approximately 2 years (January 2017 to December 2019)
  Overall survival indicator was defined as all cause death recorded at the hospital (MSO, HAD, SSR). Patients were censored at the date of last hospitalization observed (MSO/HAD/SSR/ACE).
Time to next treatment (TTNT) analysis: number of events | through study completion, approximately 2 years (January 2017 to December 2019)
  Time to next treatment indicator was defined as the time between CAR-T injection and the date of the hospitalization or palliative care.
Time to next treatment (TTNT) or death analysis: number of events | through study completion, approximately 2 years (January 2017 to December 2019)
  Time to next treatment or death indicator was defined as the first event occurring between TNTT or death presented during the hospitalization or palliative care.
Follow-up time between the CAR-T injection and the last hospital stay observed | through study completion, approximately 2 years (January 2017 to December 2019)
  Follow-up is the time between the CAR-T injection (index date) and the last hospital stay observed.
Overall cost for CAR-T hospitalization | through study completion, approximately 2 years (January 2017 to December 2019)
  The CAR-T hospitalization included Medical, Surgical, Obstetrics (MSO) hospitalization tariff and extra tariff linked to CAR-T treatment reimbursed by the health care insurance

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, East Hanover, New Jersey, United States

REFERENCES:
- See also: Results for CCTL019A0FR02 from the Novartis Clinical Trials Results Database — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17923